CLINICAL TRIAL: NCT02176603
Title: Observational, Investigator Initiated, Monocentric Study of the Endothelial Dysfunction in Adolescent and Adult Patients With Phenylketonuria Due to Phenylalanine Hydroxylase Deficiency
Brief Title: Observational Study of Endothelial Dysfunction in Phenylketonuria
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Uwe Querfeld, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: PKU-EnDys
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Phenylketonuria; Endothelial Dysfunction
Keywords: phenylketonuria, endothelial dysfunction, CKD
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine will be retained. All blood samples will be destroyed immediately after having analyzed the above mentioned parameters.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Phenylketonuria: Patients with Phenylketonuria due to phenylalanine hydroxylase deficiency
- Control group: Control group of healthy volunteers

SUMMARY:
The purpose of this study is to determine whether adolescent and adult patients with phenylketonuria who are on long-term phenylalanine-restricted diet suffer from endothelial dysfunction.

DETAILED DESCRIPTION:
The aim of the study is the examination of endothelial dysfunction and oxidative stress markers in adolescent and adult patients with phenylketonuria (PKU), in correlation to phenylalanine values und phenylalanine-restricted diet. 25-50 patients with PKU aged ≥16 years of age and a control group of 25 age- and sex-matched healthy volunteers will be included in the study.

Endothelial dysfunction will be measured by venous occlusion plethysmography on the lower legs in the PKU patients and in the control group. Wave velocity, aortic stiffness, and intima media thickness of the common carotid artery will be measured by vicorder and duplex ultrasound scanner in the PKU patients and in the control group. Analyses of phenylalanine metabolites and renal function will be performed only in the PKU patients, analyses of oxidative stress markers in the PKU patients and in the control group. Dietary protocols of the patients with PKU will be calculated for their daily phenylalanine, total protein, and calorie intake. Results of the study will be kept in the medical records and paper case report forms. Data will be analyzed only in pseudonymized form.

ELIGIBILITY:
Inclusion Criteria:

* phenylketonuria due to phenylalanine hydroxylase deficiency
* age ≥16 years

Exclusion Criteria:

* age <16 years
* pregnancy or maternity
* late-treated phenylketonuria
* phenylketonuria due a defect in BH4 synthesis or BH4 regeneration

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged ≥ 16 years with PKU diagnosed by newborn screening who are followed up in the Metabolic Unit of the Charité University Medical Center Berlin (Interdisciplinary Center for Metabolic Diseases, Dept. of Hepatology and Gastroenterology, as well as Dept. of Pediatric Endocrinology, Gastroenterology and Metabolic Diseases).
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07-22 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Post-ischaemic venous flow (measured in ml/min) in patients with PKU compared to healthy volunteers | 18 months

SECONDARY OUTCOMES:
Aortic pulse wave velocity in patients with PKU compared to healthy volunteers. Intima media thickness in patients with PKU compared to healthy volunteers. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Julia B Hennermann, MD, Principal Investigator — Johannes Gutenberg University Mainz, Germany; Uwe Querfeld, MD, Principal Investigator — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briese S, Claus M, Querfeld U. Arterial stiffness in children after renal transplantation. Pediatr Nephrol. 2008 Dec;23(12):2241-5. doi: 10.1007/s00467-008-0894-y. Epub 2008 Jun 27. PMID 18584211
- [Background] Ribas GS, Sitta A, Wajner M, Vargas CR. Oxidative stress in phenylketonuria: what is the evidence? Cell Mol Neurobiol. 2011 Jul;31(5):653-62. doi: 10.1007/s10571-011-9693-2. Epub 2011 Apr 23. PMID 21516352
- [Background] Kracht D, Shroff R, Baig S, Doyon A, Jacobi C, Zeller R, Querfeld U, Schaefer F, Wuhl E, Schmidt BM, Melk A; 4C Study Consortium. Validating a new oscillometric device for aortic pulse wave velocity measurements in children and adolescents. Am J Hypertens. 2011 Dec;24(12):1294-9. doi: 10.1038/ajh.2011.147. Epub 2011 Aug 25. PMID 21866186
- [Background] Hennermann JB, Roloff S, Gellermann J, Vollmer I, Windt E, Vetter B, Plockinger U, Monch E, Querfeld U. Chronic kidney disease in adolescent and adult patients with phenylketonuria. J Inherit Metab Dis. 2013 Sep;36(5):747-56. doi: 10.1007/s10545-012-9548-0. Epub 2012 Nov 9. PMID 23138985
- [Background] Hennermann JB, Querfeld U. Unknown pathomechanisms of renal impairment in PKU. J Inherit Metab Dis. 2013 Nov;36(6):1087-8. doi: 10.1007/s10545-013-9652-9. Epub 2013 Sep 17. No abstract available. PMID 24043382